CLINICAL TRIAL: NCT01702740
Title: A Phase 1, Double-blind, Placebo-controlled, Multiple Intravenous, Ascending-Dose Study of CNTO 136 to Evaluate Safety and Pharmacokinetics in Subjects With Cutaneous Lupus Erythematosus and to Evaluate Safety and Pharmacokinetics in a Cohort of Subjects With Systemic Lupus Erythematosus
Brief Title: A Study of the Safety and Pharmacokinetics of CNTO 136 in Patients With Cutaneous Lupus Erythematosus and Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor Research & Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013000; C0136T03 (Other: Centocor Research & Development, Inc., PA, USA); 2006-002432-25 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-10-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic
Keywords: Cutaneous lupus erythematosus; Systemic lupus erythematosus; Lupus erythematosus; Human anti-IL 6 monoclonal antibody; Sirukumab
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic | interventions — sirukumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A, 1 mg/kg CNTO 136 (Experimental)
  Interventions: Drug: 1 mg/kg CNTO 136
- Part A, 4 mg/kg CNTO 136 (Experimental)
  Interventions: Drug: 4 mg/kg CNTO 136
- Part A, 10 mg/kg CNTO 136 (Experimental)
  Interventions: Drug: 10 mg/kg CNTO 136
- Part B, 10 mg/kg CNTO 136/placebo (Experimental)
  Interventions: Drug: 10 mg/kg CNTO 136; Drug: Placebo

INTERVENTIONS:
Drug: 1 mg/kg CNTO 136 — Type=exact number, unit=mg, number=1, form=powder for solution for infusion, route=intravenous use, every 2 weeks for 6 weeks.
  Arms: Part A, 1 mg/kg CNTO 136
Drug: 4 mg/kg CNTO 136 — Type=exact number, unit=mg, number=4, form=powder for solution for infusion, route=intravenous use, every 2 weeks for 6 weeks.
  Arms: Part A, 4 mg/kg CNTO 136
Drug: 10 mg/kg CNTO 136 — Type=exact number, unit=mg, number=10, form=powder for solution for infusion, route=intravenous use, every 2 weeks for 6 weeks.
  Arms: Part A, 10 mg/kg CNTO 136; Part B, 10 mg/kg CNTO 136/placebo
Drug: Placebo — Form=liquid for infusion, route=intravenous use, every 2 weeks for 6 weeks.
  Arms: Part B, 10 mg/kg CNTO 136/placebo

SUMMARY:
The main purpose of this study was to evaluate the safety and pharmacokinetics (PK, the action of a drug in the body over a period of time) of multiple intravenous (IV) administrations of CNTO 136 in patients with cutaneous lupus erythematosus (CLE) and systemic lupus erythematosus (SLE). The secondary goal of this study was to assess the pharmacodynamics (biochemical and physiological effects of a drug and the mechanisms of action), immune response, and clinical response.

DETAILED DESCRIPTION:
In Part A of this study, patients with CLE were randomly assigned (like flipping a coin) to receive multiple IV doses of CNTO 136, a human anti-IL 6 monoclonal antibody (an immune protein that binds to interleukin 6) or placebo (a substance that appears identical to the treatment and has no active ingredients). Patients and study personnel did not know the identity of the administered treatments (double-blind study). Increasing doses were given, based on safety data collected during the initial weeks of treatment. In Part B, which was also double-blind, patients with SLE were randomly assigned to receive multiple IV doses of the highest well-tolerated dose, as determined in Part A, of CNTO 136, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cutaneous lupus erythematosus (CLE, including subacute cutaneous lupus erythematosus, discoid lupus erythematosus, or lupus erythematosus tumidus) or systemic lupus erythematosus (SLE)

  * Had a body weight less than or equal to 100 kg
  * Patients in Part A who were taking systemic medications for CLE had to be on a stable dose for 4 weeks before the first study agent infusion
  * Patients in Part B taking systemic medications for SLE had to be on a stable dose for at least 3 months before the first study agent infusion
  * Given informed consent and willing and able to adhere to the study visit schedule and other protocol requirements; agreed to avoid alcohol intake; and took adequate measures to prevent pregnancy

Exclusion Criteria:

* Significant history of or concurrent medical condition (other than lupus)
* Use of specific previous or concurrent medications or investigational therapies
* Known or suspected allergy to the study agent or it constituents, having recently donated blood, or having any significant laboratory test values requiring intervention
* Patients with SLE in Part B could not have active central nervous system lupus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 26 weeks
Pharmacokinetic profile of CNTO 136 | Up to 22 weeks
  Blood serum concentration over time
Physical examinations | Up to 26 weeks
  Assessment of head, eyes, ears, nose and throat, skin and neck, lungs, heart, abdomen, extremities, general neurologic status, and oral examination
Electrocardiograms (ECGs) | Up to 26 weeks
Sitting blood pressure | Up to 26 weeks
Heart rate | Up to 26 weeks
Respiration rate | Up to 26 weeks
Oral temperature | Up to 26 weeks
Hemoglobin | Up to 26 weeks
Hematocrit | Up to 26 weeks
Platelets and total white blood cells (WBC) | Up to 26 weeks
Albumin and total protein | Up to 26 weeks
Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) | Up to 26 weeks
Blood urea nitrogen (BUN), calcium, creatinine, and total bilirubin | Up to 26 weeks
Chloride, potassium, and sodium | Up to 26 weeks
Bicarbonate | Up to 26 weeks
Creatine kinase | Up to 26 weeks
Gamma-glutamyl-transferase | Up to 26 weeks
Glucose | Up to 26 weeks
Lymphocytes and neutrophils | Up to 26 weeks
Inorganic phosphate | Up to 26 weeks
Fasting Lipid Panel | Up to 8 weeks
  Total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), very low-density lipoprotein (VLDL), and triglycerides.

SECONDARY OUTCOMES:
Pharmacodynamics evaluations | Up to 22 weeks
  Percentage change from baseline in serum and plasma biomarker data
Immune response | Up to 22 weeks
  The formation of antibodies to CNTO 136
Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) | Up to 22 weeks
  Measurement of disease activity, scored from 0 (absent) to 70 (severe), and damage, scored from 0 (absent) to 56 (severe)
British Isles Lupus Assessment Group (BILAG) score | Up to 22 weeks
  Measures the need for alterations or intensification of therapy. The assessing physician considers each item as to its presence in the past month, and answers 0 = not present, 1 = improving; 2 = same; 3 = worse; or 4 = new.
SELENA-SLEDAI Flare Composite | Up to 22 weeks
  Assesses the presence and severity of lupus flare. Scores range from 0 (mild) to 105 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Research & Development, Inc., PA, USA Clinical Trial, Study Director — Centocor Research & Development, Inc.

REFERENCES:
- [Derived] Szepietowski JC, Nilganuwong S, Wozniacka A, Kuhn A, Nyberg F, van Vollenhoven RF, Bengtsson AA, Reich A, de Vries DE, van Hartingsveldt B, Robinson DW Jr, Gordon R, Hsu B. Phase I, randomized, double-blind, placebo-controlled, multiple intravenous, dose-ascending study of sirukumab in cutaneous or systemic lupus erythematosus. Arthritis Rheum. 2013 Oct;65(10):2661-71. doi: 10.1002/art.38091. PMID 23896980